CLINICAL TRIAL: NCT06693882
Title: Electrical Stimulation of the Optic Nerve in Patients With Glaucoma : Prospective Analysis of Perimetric Data up to 12 Months After Neuromodulatory Treatment.
Brief Title: Electrical Stimulation of the Optic Nerve in Patients With Glaucoma.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Glaucoma Center of San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00080468
Record Dates: First submitted 2024-11-15; First posted 2024-11-18 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Intervention Model Description: Prospective analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with glaucoma undergoing electrical stimulation of the optic nerve (Other): Single arm study of patients with glaucoma undergoing electrical stimulation of the optic nerve
  Interventions: Device: EYETRONIC Nextwave System

INTERVENTIONS:
Device: EYETRONIC Nextwave System — Eyetronic Nextwave is a neurostimulation device that stimulates the optic nerve non-invasively using transcranial alternating current stimulation delivered through goggles in patients presenting with glaucoma.
  Eyetronic is approved in Europe for the treatment of glaucoma to possibly delay progression of visual field (VF) loss for at least 12 months. The indication for use in Europe includes all patients suffering from neuropathies of the optic nerve resulting in loss of VF. Two studies conducted in Europe have demonstrated improvement in visual fields following 10-days of optic nerve stimulation treatment with this device. In the current study, the Eyetronic system will be used to treat only those individuals who have visual field loss from glaucoma.

SUMMARY:
The goal of this observational study is to evaluate electrical stimulation of the optic nerve with the Eyetronic Nextwave System device as a possible treatment for glaucoma.

The main question it aims to answer is:

Could this therapy be an option to counteract the loss of visual field seen in glaucoma and thus delay the progression of the disease?

Participants will have approximately 14-18 study visits during 12 months including 10 visits for the electrical stimulation treatment. The treatment involves electrically stimulating the optic nerve by an external approach via the facial skin.

DETAILED DESCRIPTION:
1. During the study visits participants will have: general eye examination (visual acuity check, examination of the front and back of the eye, eye pressure measurement, pupil dilation), Visual field (VF) testing, Imaging the optic nerve with Optical Coherence Tomography (OCT), Optic nerve photos.
2. The treatment will include ten sessions during 2 weeks on an outpatient basis in a quiet and dimly lit room with the patient comfortably seated or lying down in a reclining chair. Each treatment session will last approximately 60 minutes including the time to determine the treatment settings.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years or older who have glaucoma
* Humphrey visual field mean deviation (MD) values between - 6 dB and -20 dB

Exclusion Criteria:

* Age < 18 years
* Implanted electronic devices
* Metallic artifacts in the head (except dentures)
* Migraine
* Epilepsy
* Brain tumor
* Pregnancy
* Breastfeeding patients
* Uncontrolled intraocular pressure (IOP)
* IOP lowering medication started less than six months before enrollment
* Any intraocular surgery less than 6 months before enrollment
* Arterial hypertension without appropriate treatment
* Acute retinal hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in visual field mean deviation (MD) from baseline to post-treatment | 12 months
  Visual field testing will be performed with the Humphrey field analyzer (Carl Zeiss Meditec)

SECONDARY OUTCOMES:
Change in retinal nerve fiber layer (RNFL) thickness from baseline to post-treatment | 12 months
  Optical coherence tomography (OCT) will be performed with the Cirrus OCT device (Carl Zeiss Meditec)

CONTACTS AND LOCATIONS:
Locations (1):
- Glaucoma Center of San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No